CLINICAL TRIAL: NCT00681369
Title: Observational Usage Study of Faslodex in Patients Suffering From Initial Breast Cancer in France
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar - Medical Science Director, AstraZeneca
Other Study IDs: NIS-OFR-FAS-2007/1
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; fulvestrant; longitudinal study; France
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients suffering from initial breast cancer, treated with Faslodex, treatment which was stopped during 2007

SUMMARY:
the purpose of this study is to describe the way Faslodex is used in France, in patients suffering from initial breast cancer, that is to evaluate Faslodex treatment duration and to determine patients profile

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from initial breast cancer, treated with Faslodex, treatment which was stopped during 2007

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital sample
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2007-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluate Faslodex therapeutic strategy and treatment duration | At the end of the study
Describe the characteristics of patients treated with Faslodex | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alain FLINOIS, Principal Investigator — TNS Healthcare - France138, avenue Marx Dormoy92120 Montrouge